CLINICAL TRIAL: NCT04125173
Title: The Effect of Lower Pneumoperitoneum Pressure During Laparoscopic and Robotic Hysterectomy: A Randomized Controlled Trial
Brief Title: Effect of Lower Pneumoperitoneum Pressure During Laparoscopic and Robotic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Rachael Bailey Smith, Rachael Smith, DO Fellow Minimally Invasive Gynecology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1909975965
Record Dates: First submitted 2019-07-29; First posted 2019-10-14 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Hysterectomy; Pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Three arms including those with pneumoperitoneum pressure of 15mmgHg versus 12mmgHg vs 10 mmHg during laparoscopic or robotic hysterectomy for benign indications.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research coordinator will have randomized the patient into one of the 3 arms. The randomized pneumoperitoneum pressure will be set for the surgical procedure and blinded to the surgeon and first assistant, either fellow or resident.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Pneumoperitoneum pressure = 15mmHg (Active Comparator): 1. Pneumoperitoneum will be set at 15mmHg
  Interventions: Other: Pneumoperitoneum pressure = 15mmHg
- 2. Pneumoperitoneum pressure = 12mmHg (Active Comparator): 2.Pneumoperitoneum will be set at 12mmHg
  Interventions: Other: Pneumoperitoneum pressure = 12mm Hg
- 3. Pneumoperitoneum set at 10mmHg (Active Comparator): 3. Pneumoperitoneum will be set at 10mmHg
  Interventions: Other: Pneumoperitoneum pressure = 10mmHg

INTERVENTIONS:
Other: Pneumoperitoneum pressure = 15mmHg — Randomized pneumoperitoneum 1
  Arms: 1. Pneumoperitoneum pressure = 15mmHg
Other: Pneumoperitoneum pressure = 12mm Hg — Randomized pneumoperitoneum 2
  Arms: 2. Pneumoperitoneum pressure = 12mmHg
Other: Pneumoperitoneum pressure = 10mmHg — Randomized pneumoperitoneum 3
  Arms: 3. Pneumoperitoneum set at 10mmHg

SUMMARY:
With the limited evidence that lower pneumoperitoneum pressures improve postoperative pain in laparoscopic or robotic hysterectomy for benign indications, we would like to determine if we can both further validate this idea but also show that it has minimal effect on physician satisfaction performing the surgery.

DETAILED DESCRIPTION:
Minimally invasive hysterectomy, including conventional laparoscopic and robotic-assisted hysterectomy, is a commonly performed gynecologic surgery that universally results in postoperative pain for patients. Opioid medications are helpful to control postoperative pain and are routinely given to women who undergo minimally invasive hysterectomy. However, opioid abuse is on the rise in the United States, and there is increased awareness of misuse leading to abuse, overdose, and chronic opioid use. In addition to narcotic usage, postoperative pain also has negative effects on patient satisfaction and length of stay in the post-anesthesia care unit (PACU) leading to potential hospital admission. There is existing evidence that reducing the pressure used to create the pneumoperitoneum during laparoscopic surgery may affect pain scores that patients endorse in the PACU. Due to improved postoperative pain, patients may have decreased opioid use in the PACU and at home, shorter hospital stay, and improved overall patient satisfaction. If lower pneumoperitoneum pressures during laparoscopic surgery can be shown to reduce postoperative pain, then the ultimate question becomes whether there is ability to adapt this practice of using lower pressures to maintain pneumoperitoneum. It is unclear whether physician satisfaction will be affected.

There are several publications investigating the effect of lower pneumoperitoneum pressures on postoperative pain. A systematic review in 2016 included 238 patients (three RCTs), showed pneumoperitoneum pressures of 8mmHg had a statistically significant although minimal decrease in postoperative pain compared to 12mmHg, although lower pressures were associated with worse visualization. The authors concluded that the systematic review was inconclusive and further studies were necessary. A randomized pilot study with 60 patients comparing low pressure (7mmHg) using the AirSeal System versus standard insufflation (15mmHg), showed lower postoperative shoulder pain in the group with lower pressure using the AirSeal system. Two abstracts in the Journal of Minimally Invasive Gynecology present retrospective studies showing decreased postoperative pain with lower pneumoperitoneum pressure. The first abstract is from 2015, included a sample size of 170 patients who underwent benign robotic gynecologic surgery, 85 patients in each arm (12mmHg and 15mmHg). They showed no difference in median recovery time in the PACU and significantly lower median first pain score (5 vs 6, p=.04). The second abstract is from 2018 and included a sample size of 598 patients who underwent benign robotic gynecologic surgery, 99 patients in 15mmHg arm, 100 patients in 12mmHg arm, 99 patients in 10mmHg arm, and 300 patients in 8mmHg arm. They showed lower initial pain scores with each degree of lower pressure (5.9 vs 5.4 vs 4.4 vs 3.8, p=<.0001) and shorter hospital stays with lower pressures. They showed no difference in operative times or blood loss in the four arms. Similar studies have been done with cholecystectomy patients that have shown improved postoperative shoulder pain with lower pneumoperitoneum pressures. There is also an ongoing clinical trial that is still recruiting patients that is studying this similar comparison using 9mmHg vs 15mmHg with and without the AirSeal system.

However, the literature summarized here has never included blinding the intervention of lower pneumoperitoneum pressure to the surgeon to determine awareness of pressure and its effect on visualization and physician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* greater than or equal to 18 years old
* English-speaking
* undergoing laparoscopic or robotic total hysterectomy for benign indications by one of the two minimally invasive gynecologic surgeons at Banner University Medical Center - Phoenix

Exclusion Criteria:

* patients with body max index >35
* American Society of Anesthesiologists (ASA) score III or IV
* preoperative uterine weight estimated to be greater than 500gm (measured by sonography and using the following formula: length x width x anteroposterior diameter x 0.52)
* patients on chronic opioids for chronic pain (defined as > 3 months regular opioid use)
* patients who refuse participation in the study
* patients who do not provide informed consent

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Physician Satisfaction Part 1 | From completion of surgery to one hour postoperative
  Physician satisfaction questionnaire completed immediately postoperative, 3 questions in length and measured with VAS score (0-5)
Physician Satisfaction Part 2 | From completion of surgery to one hour postoperative
  Included in the physician satisfaction questionnaire is presumed pneumoperitoneum pressure, measured as 10mmHg, 12mmHg, or 15mmHg (circle one - 10mmHg, 12mmHg, 15mmHg)
Physician Satisfaction Part 3 | From completion of surgery to one hour postoperative
  Included in the physician satisfaction questionnaire are two yes/no questions on effect of pneumoperitoneum on visualization and operative time (circle one - yes, no)

SECONDARY OUTCOMES:
Postoperative Pain | From completion of surgery to 24 hours postoperative
  Self reported pain intensity in PACU (VAS 0-10) first reported and maximum pain score, pain score at 6 hours postoperative, and pain score at 24 hours postoperative
Postoperative Shoulder Pain | From completion of surgery to 24 hours postoperative
  Self reported shoulder pain intensity (VAS 0-10) at 6 hours postoperative and pain score at 24 hours postoperative

OTHER OUTCOMES:
Narcotic usage | From completion of surgery to 24 hours postoperative
  Morphine equivalent units in PACU and at 24 hours postoperative
Length of hospital stay | From completion of surgery to hospital discharge time up to 7 days
  Time in minutes of length of stay in hospital
Patient Satisfaction | From completion of surgery to 24 hours postoperative
  Patient satisfaction questionnaire completed 24 hours postoperative over the phone, 2 questions in length, VAS score (0-5) on satisfaction with overall postoperative pain and shoulder postoperative pain
Intraoperative Respiratory Parameters: Peak inspiratory pressure | From start of surgery to end of surgery
  Peak inspiratory pressure
Intraoperative Respiratory Parameters: Tidal volume | From start of surgery to end of surgery
  Tidal volume
Intraoperative Respiratory Parameters: End tidal CO2 | From start of surgery to end of surgery
  End tidal CO2

CONTACTS AND LOCATIONS:
Overall Officials: Michael Foley, MD, Study Chair — Banner University Medical Center
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identifed individual participant data for all primary and secondary outcomes measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requesters will be required to sign a data access agreement.

REFERENCES:
- [Background] Kyle EB, Maheux-Lacroix S, Boutin A, Laberge PY, Lemyre M. Low vs Standard Pressures in Gynecologic Laparoscopy: a Systematic Review. JSLS. 2016 Jan-Mar;20(1):e2015.00113. doi: 10.4293/JSLS.2015.00113. PMID 26955258
- [Background] Bogani G, Uccella S, Cromi A, Serati M, Casarin J, Pinelli C, Ghezzi F. Low vs standard pneumoperitoneum pressure during laparoscopic hysterectomy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):466-71. doi: 10.1016/j.jmig.2013.12.091. Epub 2013 Dec 25. PMID 24374246
- [Background] Sroussi J, Elies A, Rigouzzo A, Louvet N, Mezzadri M, Fazel A, Benifla JL. Low pressure gynecological laparoscopy (7mmHg) with AirSeal(R) System versus a standard insufflation (15mmHg): A pilot study in 60 patients. J Gynecol Obstet Hum Reprod. 2017 Feb;46(2):155-158. doi: 10.1016/j.jogoh.2016.09.003. Epub 2017 Jan 30. PMID 28403972
- [Background] 3. Kim DK, Cheong ILY, Lee GY, Cho JH. Low pressure (8 mm Hg) pneumoperitoneum does not reduce the incidence and severity of postoperative nausea and vomiting (PONV) following gynecologic laparoscopy. Korean J Anesthesiol. 2006.
- [Background] Topcu HO, Cavkaytar S, Kokanali K, Guzel AI, Islimye M, Doganay M. A prospective randomized trial of postoperative pain following different insufflation pressures during gynecologic laparoscopy. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:81-5. doi: 10.1016/j.ejogrb.2014.09.003. Epub 2014 Sep 16. PMID 25265495
- [Background] Nasajiyan N, Javaherfourosh F, Ghomeishi A, Akhondzadeh R, Pazyar F, Hamoonpou N. Comparison of low and standard pressure gas injection at abdominal cavity on postoperative nausea and vomiting in laparoscopic cholecystectomy. Pak J Med Sci. 2014 Sep;30(5):1083-7. doi: 10.12669/pjms.305.5010. PMID 25225531